CLINICAL TRIAL: NCT04758741
Title: Investigating the Impact of Acceptance and Commitment Therapy on Resiliency in Women Affected by Domestic Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatemeh Khakshoor (Other)
Responsible Party: Sponsor-Investigator, Fatemeh Khakshoor, Investigator, Arak University of Medical Sciences
Organization: Arak University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.ARAKMU.REC.1399.226
Record Dates: First submitted 2021-01-25; First posted 2021-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Domestic Violence
Keywords: Acceptance and commitment therapy; Resiliency; Domestic violence
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Individuals are randomly divided into two groups: intervention (n = 40) and control (n = 40). The members of the intervention group in groups of 10 will receive acceptance and commitment treatment in 8 90-minute sessions once a week according to Hayes (2006) approach in Mashhad Al-Koubeh Health Center by a consultant (researcher) trained. The control group also receives 8 counseling sessions per week by the same "Health Education" consultant in groups of 10 in the same center. One week after the end of the eighth session and one month later, the questionnaires are completed again by trained questioners for both groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sequencing will be centralized in such a way that the list of random allocation sequences is provided to someone outside the research team. As soon as a person is eligible to participate in the study, the sampler contacts the person who has the random assignment sequence and he or she, according to the sequence list, gives the code to the participants to enter the study. Acceptance and commitment therapy sessions are held by a trained researcher. At the evaluation stage, one week and one month after the intervention, the questionnaires are completed by trained questioners. The statistical consultant who will assist in the data analysis will be unaware of the codes of the participants in the groups. Therefore, the study will be of the three-blind type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and commitment treatment (Experimental): The members of the intervention group receive one session of acceptance and commitment treatment per week according to Hayes (2006) approach in groups of 10 in 8 sessions of 90 minutes by a trained counselor (researcher) in Mashhadalkoubeh Health Center.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Health Education (Sham Comparator): This rct has one arm and health education is done only for the purpose of blinding the study so that the participant does not know which of the control or intervention groups it is in and has no comparative aspect and has nothing to do with resilience.
  Interventions: Other: placebo

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Investigating the impact of Acceptance and Commitment Therapy on Resiliency in women affected by domestic violence
  Arms: Acceptance and commitment treatment
Other: placebo — This rct has one arm and health education is done only for the purpose of blinding the study so that the participant does not know which of the control or intervention groups it is in and has no comparative aspect and has nothing to do with resilience
  Arms: Health Education

SUMMARY:
This study is a randomized controlled counseling intervention with pre-test, post-test and control groups. After obtaining informed consent from 80 women affected by domestic violence that referred to the health centers of the villages covered by Al-Kooh Mashhad Health Center (Mashhad Al-Kooh Health Center, Michan, Mosleh Abad) and Mashhad Al-Kobeh Health Center, and are eligible to enter Rct are. A woman who has been subjected to domestic violence is someone who has obtained at least one score on the (cts2) questionnaire .

Then, these people are randomly divided into two groups of intervention (n = 40) and control (n = 40). The members of the intervention group in groups of 10 are treated in 8 sessions of 90 minutes once a week based on "acceptance and commitment treatment" based on Hayes (2006) approach by a trained consultant (researcher) in Mashhad AL-koubeh Health Center. The control group also receives 8 counseling sessions once a week by the same "health education" consultant in groups of 10 at the same center. One week after the end of the eighth session and one month later, the questionnaires are completed again by trained questioners for both groups.

The instruments studied in this study include demographic questionnaire, conflict resolution tactics questionnaire (cts 2) and resilience questionnaire (Connor-Davidson). Data analysis is performed using descriptive and inferential statistics with SPSS software version 23.

DETAILED DESCRIPTION:
Sampling:

In this project, (80 people) eligible women (with at least one score from the CTS2 questionnaire) are selected through available health centers in the villages covered by Mashhad-e-Kobeh Health Center and Mashhad-e-Koboeh Health Center by available sampling method. They are randomly divided into intervention and control groups.

Randomization type:

Randomization is blockchain. 20 blocks with a volume of 4 are used, two allocations for the control group and two allocations for the intervention group. Random sequencing is done using a web-based random site (https://www.sealedenvelope.com).

Sequence Hiding: Sequence hiding is when someone outside the research team has a random assignment list. As soon as a person is eligible to participate in the study, the sampler contacts the person who has a random assignment sequence and he / she gives the code to the participants to enter the study according to the sequence list.

Acceptance and commitment therapy sessions are held by a researcher who has learned the workshop before starting the project. In the evaluation phase, one week and one month after the intervention, the questionnaires are completed by trained questioners. The statistical consultant who will help analyze the data is unaware of the codes of the participants in the groups. Therefore, the study will be of the three-blind type.

Data collection method:

Questionnaires are completed by pre-intervention interviews by trained researchers and samplers and in the evaluation phase after the intervention and follow-up by trained interviewers. Before starting the study, questioners with high public and social relations are selected for sampling and during a session, the necessary training is given to them by the researcher. During the briefing, the objectives of the study and the work process, the sampling method, the confidentiality of customer information and the privacy of the participant, and all ethical principles related to domestic violence research are taught to the samplers.

Data collection tools:

The instruments studied in this study include Demographic Questionnaire, CTS2 Conflict Resolution Tactics Questionnaire (to determine the status of violence) and Connor and Davidson Resilience Questionnaire (to determine the status of resilience).

Hypothesis:

Acceptance and commitment to therapy affect women's resilience to domestic violence.

all purpose: The effect of treatment acceptance and commitment on the resilience of women affected by domestic violence is determined.

Specific objectives:

Determining and comparing the mean resilience score in the intervention and control groups, before, one week after the intervention and one month after the intervention.

Functional purpose:

If the effectiveness of acceptance and commitment therapy in improving the resilience of women affected by domestic violence is confirmed, this intervention method can be used in counseling centers and its use can be taught to service providers, especially midwives. Applying this method will probably be effective in reducing the rate of violence and mutual violence against women, promoting women's health, improving marital relations and marital satisfaction, strengthening the family and reducing the rate of divorce.

ELIGIBILITY:
Inclusion Criteria:

* Giving informed written consent.
* Having experience of domestic violence by the husband for at least the last six months (obtaining at least one grade from the aggressive form of the cts2 questionnaire).
* Ability to speak Persian.
* Having at least a third grade of secondary education (to Reason for being able to understand the concepts related to intervention and being able to do homework)
* Being Iranian.
* Being married.
* Not being pregnant during pregnancy and postpartum (up to 6 months postpartum).
* Not taking psychedelic, anti-anxiety and anti-depressant drugs In the interval of 6 months before participating in the study and during the study.
* No consciousness disorder.
* No history of hospitalization in the psychiatric ward.
* No incurable physical disease such as cancer Or malignant tumors.
* Not experiencing any severe stress such as divorce, accident, bereavement of relatives in the last six months.
* No simultaneous participation in counseling courses with content similar to the present intervention.

Exclusion Criteria:

* Not participating in two or more treatment sessions.
* Experiencing any severe stress during the study, such as incurable physical illness such as cancer or malignant tumors, pregnancy during the study, divorce, accident, bereavement of relatives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Having experience of domestic violence by the husband for at least the last year.
Enrollment: 80 (Actual)
Dates: Start 2020-11-28 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
change of Resiliency | from before the intervention to one week and one month after the intervention
  Resilience refers to a person's score on the Connor & Davidson (2003) Questionnaire (CD-RISC).The minimum score on this scale is zero and the maximum score is 100. A higher score indicates more resilience, meaning a better situation.

SECONDARY OUTCOMES:
Change in the experience of domestic violence | from before the intervention to one month after the intervention
  A violence woman is a woman who has answered at least one question from the (cts2) questionnaire.The minimum score on this scale is zero and the maximum score is 432. A higher score indicates more experience of violence and a worse situation.

CONTACTS AND LOCATIONS:
Overall Officials: abed majidi, phd, Study Chair; azam moslemi, phd, Study Chair — Arak University of Medical Sciences; sakineh taherkhani, phd, Principal Investigator — Arak University of Medical Sciences
Locations (1):
- Mashhad Alkoubeh Health Center, Arak, Markazi Province, Iran

IPD SHARING:
Plan to Share IPD: No